CLINICAL TRIAL: NCT00293124
Title: An Open-label Trial of Glivec in Patients With Unresectable or Metastatic Malignant Gastrointestinal Stromal Tumors Expressing C-kit.
Brief Title: Open-label Trial of GlivecWith Unresectable or Metastatic Malignant Gastrointestinal Stromal Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/GIST 1.2.001; CSTI571BIC07
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2012-05

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; Glivec
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Glivec — 400mg p.o./day in a population of patients with locally advanced (=not amenable to surgery with curative intent) or metastatic malignant GIST. Glivec® may be increased to 600 mg p.o./day and then 800 mg p.o./day (400 mg b.i.d.) if the patient is progressing

SUMMARY:
The rationale is to assess the clinical and biological activity of Imatinib and to compare the data with historic data.

Additionally this study has been designed to gain more experience with the treatment of GIST in several Central and Eastern European Countries.

DETAILED DESCRIPTION:
This is a multicenter open label clinical trial to be performed in patients with incurable malignant GISTs that are unresectable or metastatic. Approximately 150 patients will enter the trial.

Patients will receive Imatinib 400 mg p.o./day for a period of up to 24 months provided that in the opinion of the investigator the patient is benefiting from treatment with Imatinib, and in the absence of any safety concerns.

Treatment after completion of the 24 months study is at the discretion of the investigator. Imatinib should be increased to 600 mg p.o./day and then to 400 mg b.i.d if the patient is progressing on the respective dose level.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years of age
* Histologically documented diagnosis of GIST which is malignant as well as unresectable (=not amenable to surgery with curative intent) and/or metastatic and therefore incurable Immunohistochemical documentation of c-kit (CD117) expression by tumor
* At least one measurable site of disease (as defined by Southwestern Oncology Group Solid Tumor Response Criteria) which has not been previously embolised or irradiated
* Performance status 0,1, 2 or 3 (ECOG)
* Adequate end organ function, defined as the following: total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 x UNL (or < 5 x ULN if hepatic metastases are present), creatinine < 1.5 x ULN, ANC > 1.5 x 109/L, platelets > 100 x 109/L
* Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* Life expectancy of at least 6 months
* Written, voluntary, informed consent
* Patients who were previously treated with chemotherapy will be eligible for this study
* Patient who are at least 5 years free of melanoma will be eligible for this study

Exclusion Criteria:

* Patient has received any other investigational agents within 28 days of first day of study drug dosing
* Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention and CECOGs' approval is obtained, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed
* Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e., congestive heart failure, myocardial infarction within 6 months of study)
* Female patients who are pregnant or breast-feeding.
* Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection)
* Patient has a known brain metastasis
* Patient has an acute or known chronic liver disease (i.e., chronic active hepatitis, cirrhosis)
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection
* Patient received chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin-C) prior to study entry
* Patient previously received radiotherapy to >= 25 % of the bone marrow
* Patient had a major surgery within 2 weeks prior to study entry
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent
* Therapeutic anticoagulation with warfarin (e.g. Coumadin® or Coumadine®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2004-03; Primary Completion 2006-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Time to Disease Progression | until PD

SECONDARY OUTCOMES:
Time to Disease Progression | until PD
Overall Survival | until death

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brodowicz, MD, Principal Investigator — University Clinic of Internal Medicine I / Clinical Oncology
Locations (16):
- AKH, Universitätsklinik für Innere Medizin 1, Vienna, Austria
- Institute of Oncology Sarajevo, Sarajevo, Bosnia and Herzegovina
- Bulgaria (3):
  - SBALO National Oncology Center, Sofia
  - National Oncological Center Hospital, Sofia
  - Sofia Cancer Center compl. Mladost ,, Sofia
- Croatia (2):
  - Clinical Hospital Split, Center of Oncology, Split
  - University Hospital Rebro, Zagreb
- Czechia (2):
  - FN Bulovka, Prague
  - Radioterapeticko-onkologicke. Oddeleni FN Motol, Prague
- Lithuanian Oncology Center,, Vilnius, Lithuania
- Romania (3):
  - Institutul Oncologic Bucuresti, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Emergency Clinical County Hospital , Clin Oncol. Dep, Craiova
- Institut za onkologiju i, Belgrade, Serbia
- National Institute of Oncology, Bratislava, Slovakia
- Oncology Institute Ljubljana, Ljubljana, Slovenia

REFERENCES:
- See also: Related Info — http://www.cecog.org